CLINICAL TRIAL: NCT02250261
Title: Socio-ecological Intervention to Promote Active Commuting to Work
Acronym: KÄPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UKK Institute (Other)
Collaborators: Tampere University of Technology (Other); Department of Transport and Streets, City of Tampere (Unknown); Ecofellows Ltd, City of Tampere (Unknown); University of Oxford (Other); University of Graz (Other)
Responsible Party: Principal Investigator, Minna Aittasalo, Senior Researcher, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 179
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Active Travel
Keywords: walking; cycling; intervention; physical activity; environment; promotion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KÄPY group (Experimental): Workplaces, which are supported to promote employees' ACW.
  Interventions: Behavioral: KÄPY
- Comparison group (No Intervention): Workplaces, which are not supported to promote employees' ACW but will be offered support to do so after the study.

INTERVENTIONS:
Behavioral: KÄPY
  Arms: KÄPY group

SUMMARY:
Background Cycling and walking to work is a natural way of increasing physical activity in a working population. However, the evidence on the effectiveness and cost savings of promoting active work commuting (ACW) is thin. This cluster-randomized, controlled study aims to promote ACW with environmental, social and behavioral strategies in two large workplace areas in Tampere, Finland. The paper de-scribes the protocol, evaluation and baseline findings of the study.

Methods The enrollment of the workplaces took place in 2014-15. In Phase 1, the impacts of environmental strategies (improvements to the walking and cycling trails) were evaluated in Area1 including 11 workplaces. In Phase 2, five more workplaces were recruited from Area2 to evaluate the impacts of social and behavioral strategies accustomed for each workplace. The workplaces in both areas were then randomized into experimental (EXP, n=6+2) and comparison group (COM, n=5+3). EXP promoted ACW with social and behavioral strategies; COM participated in data collection only but will have the same support post-intervention. The primary outcome is the change in employees' self-reported and accelerometer-based ACW. The secondary outcomes include e.g. the changes in employees' self-rated health and subjective wellbeing at work, the change in the number of walkers and cyclists based on the traffic calculations and the change in the quality of walking and cycling trails based on camera auditing (Area1 only). External validity of the intervention is as-sessed with the compliance rates of the workplaces and employees as well as with the fidelity of the environmental, social and behavioral strategies. Health Economic Assessment Tool for Cycling and Walking (HEAT) is used to assess the cost savings of the multilevel intervention. In addition, environmental variables and types that promote ACW and mediate and moderate the effects of environmental strategies are examined.

Results and discussion This study is one of the first in Finland to combine interdisciplinary collaboration between practi-tioners and researchers working in the fields of transportation, urban design, physical activity and sustainable development to promote ACW. The findings benefit all stakeholders interested in pro-moting ACW in urban context. The study will also produce supportive material for promoting ACW at the workplaces.

ELIGIBILITY:
Inclusion Criteria:

All voluntary employees in the workplaces located in the specific area

Exclusion Criteria:

No exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in self-reported means of transportation to work | 1 year
  Proportion of employees walking or cycling to work (%)
Change in self-reported weekly AWC | 1 year
  Mean number of days employees walk or cycle to work
Change in accelerometer-based daily duration of walking and cycling to work | 1 year
  Daily minutes of AWC (mean)

SECONDARY OUTCOMES:
Change in self-rated health | 1 year
  Employees self-reported health
Change in subjective well-being at work | 1 year
  Includes six indicators self-reported by the employees
Change in restrictions to ACW | 1 year
  Self-reported by the employees and grouped into four levels
Change in motivation for ACW | 1 year
  Includes six indicators self-reported by the employees
Change in injuries due to ACW | 1 year
  Self-reported by the employees
Change in the use of the main walking and cycling trail (Area1) | 1 year
  Measured with fixed-point traffic calculations
Change in the quality of the main walking and cycling trail | 1 year
  Audited by cycling the trails with GPS

OTHER OUTCOMES:
Cost-savings | 1 year
  HEAT
Cost-effectiveness | 1 year
  cost-effectiveness ratio
Environmental evaluation | 1 year
  Urban environmental variables and types
Environmental evaluation | 1 year
  Variables, which mediate and moderate the effects of environmental strategies

CONTACTS AND LOCATIONS:
Overall Officials: Minna Aittasalo, D.Sc., Principal Investigator — UKK Institute
Locations (2):
- Finland (2):
  - UKK Institute, Tampere, Pirkanmaa
  - The UKK Institute for Health Promotion Research, Tampere, Pirkanmaa

REFERENCES:
- [Result] Aittasalo M, Tiilikainen J, Tokola K, Seimelä T, Sarjala S-M, Metsäpuro P, Hynynen A, Suni J, Sievänen H, Vähä-Ypyä H, Vaismaa K, Vakkala O, Foster C, Titze S, Vasankari T. Socio-Ecological Intervention to Promote Active Commuting to Work: Protocol and Baseline Findings of a Cluster Randomized Controlled Trial in Finland. Int J Environ Res Public Health. 2017 Oct; 14(10): 1257. Published online 2017 Oct 20. doi: 10.3390/ijerph14101257
- See also: Related Info — http://www.ukkinstituutti.fi